CLINICAL TRIAL: NCT05280080
Title: Neuromuscular and Perceptual Responses, Pain Intensity and Performance During Resistance Exercise With a Self-regulated Dual-task in Patients With Severe Knee Osteoarthritis
Brief Title: Exercise With Dual Task in Knee Osteoarthritis
Acronym: DTOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, José Casaña Granell, Head of the Physiotherapy Department, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OA-22-02
Record Dates: First submitted 2022-02-15; First posted 2022-03-15 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Electromyography; Muscle Activity; Resistance Training
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular Task (Active Comparator): Knee extensions.
  Interventions: Other: Resistance exercise
- Dual Task (Experimental): Knee extensions while also doing a self-regulated mathematical dual-task.
  Interventions: Other: Resistance exercise

INTERVENTIONS:
Other: Resistance exercise — Do the maximum number of repetitions of externally-resisted (50% 1RM) knee extensions.

SUMMARY:
The purpose of this study is to evaluate the neuromuscular and perceptual responses, pain intensity and performance in patients with severe knee osteoarthritis in a preoperative setting with low-load resistance training with a self-regulated mathematical dual-task.

ELIGIBILITY:
Inclusion Criteria:

* men and women above 55 years old.
* diagnosed with severe knee osteoarthritis.
* scheduled for unilateral TKA surgery in a local hospital during 2021- 2022.

Exclusion Criteria:

* pain in the contralateral limb (maximum pain, ≥80 of 100 mm on a VAS during daily activities).
* another hip or knee joint replacement in the previous year.
* any medical condition in which exercise was contraindicated.
* participated in exercise programs (>2 days/week, training at intensities of 10-15RM) in the 6 months prior to the study.
* history of stroke, brain surgery, major depression, or any self-perceived cognitive alterations that could affect the performance of dual tasks.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Self-reported pain intensity (Visual Analogue Scale (VAS) Scale 0-10) | Pre exercise, immediate post session, and 10 minutes after session.
  Change from baseline to the end of the session, and the change between the dual-task and the regular condition.
Pressure pain thresholds | Pre exercise, immediate post session, and 10 minutes after session.
  Change from baseline to the end of the session, and the change between the dual-task and the regular condition.
HDsEMG | During each experimental session and during each exercise condition.
  Change from baseline to the end of the session, and the change between the dual-task and the regular condition.
Performance | During each experimental session and during each exercise condition.
  Maximum number of exercise repetitions performed.

SECONDARY OUTCOMES:
Tampa Scale of Kinesiophobia (TSK 11) | Pre session.
  Its score range is 11-44, with higher scores reflecting worse condition.
Pain Catastrophizing Scale (PCS) | Pre session.
  People are asked to indicate the degree to which they have certain thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale. A total score is yielded (ranging from 0-52), along with three subscale scores assessing rumination, magnification and helplessness, with higher scores reflecting worse condition.
Chronic Pain Self-Efficacy Scale (CPSS) | Pre session.
  The Chronic Pain Self-Efficacy Scale (CPSS) is designed to measure chronic pain patients' perceived self-efficacy to cope with the consequences of chronic pain. The CPSS measures three domains of pain self-efficacy: pain management, physical functioning, and coping with symptoms. A total score is yielded (ranging from 220-2200), with higher scores reflecting a better condition.
WOMAC questionaire for patients with hip or knee osteoarthritis. | Pre session.
  The WOMAC is a disease-specific self-administered questionnaire for patients with hip or knee osteoarthritis. It has a multidimensional scale made up of 24 items grouped into three dimensions: pain (5 items), stiffness (2 items) and physical function (17 items). For each item, it uses a Likert scale with five response levels, representing different degrees of intensity (none, mild, moderate, severe or extreme) that are scored from 0 to 4. The final score for the WOMAC is determined by adding the aggregate scores for pain, stiffness and function. The higher the score, the worse the patient's condition.
Heart Rate | Pre exercise, immediate post session, and 10 minutes after session.
  Change from baseline to the end of the session, and the change between the dual-task and the regular condition.
Perceived difficulty of the dual-task. | Immediate post exercise.
  Based on an 11-point numerical rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: José Casaña, Principal Investigator — University of Valencia; Joaquín Calatayud, Study Chair — University of Valencia
Locations (1):
- Clinic Universitary Hospital of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No